CLINICAL TRIAL: NCT00579683
Title: A Prospective Registry for Patients With Acquired Resistance to Small Molecule Kinase Inhibitors in Non-Small-Cell Lung Cancer
Brief Title: Registry for Patients With Acquired Resistance to Small Molecule Kinase Inhibitors in Non-Small-Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-103
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Unresectable or Metastatic Non-small Cell Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer; NSCLC; metastatic disease; resistent disease; RNA analysis; 04-103
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy material will be processed to obtain RNA for analysis of EGFR sequence. Sequencing of additional candidate genes and other studies will follow if sufficient material is available.

GROUPS / COHORTS (1):
- 1: This is a protocol to study tissue specimens to identify changes in tumor DNA in NSCLC patients who have previously responded to therapy and who have subsequently experienced disease progression.
  Interventions: Other: Tumor core biopsy for RNA isolation

INTERVENTIONS:
Other: Tumor core biopsy for RNA isolation — RNA isolation will be carried out using approximately 25 mg of gross tissue from these tumor specimens.

SUMMARY:
The purpose of this study is to try to learn more about how small molecule kinase inhibitors work in treating lung cancer. Some early studies have shown that gefitinib, erlotinib and similar drugs are more likely to work if a particular DNA change (also known as a mutation) is found in a protein that is important in lung cancer. This protein is called the epidermal growth factor receptor (EGFR). Since small molecule kinase inhibitors sometimes stop working, we would like to examine your tumor to learn why these medicines are not working as well. Your tumor will be examined for a variety of things including changes in the DNA of the EGFR. We will also sequence parts of the genes for HER2, HER3, HER4, and KRAS, other proteins thought to be important in lung cancer.

DETAILED DESCRIPTION:
The goal of this protocol is to determine mechanisms of resistance to epidermal growth factor (EGFR) tyrosine kinase inhibitors (EGFR-TKI) in non-small cell lung cancer (NSCLC). A number of trials have shown small molecule kinase inhibitors to be active agents in the treatment of NSCLC [1]. Clinically these drugs have been noted to produce dramatic but infrequent responses. Mutations in the epidermal growth factor receptor have been shown to correlate with sensitivity to gefitinib and erlotinib[2,3]. However, we know that most patients who have initial responses to EGFR-TKI eventually progress. The mechanism of acquired clinical resistance to these inhibitors in patients incompletely understood.

This is a protocol to study clinical characteristics and biopsy tissue of patients with non-small cell lung cancer who have had previous clinical response to small molecule kinase inhibitors and subsequently experience progression of disease. The tissues and other specimens will be used to carry out laboratory studies to explore the molecular basis of sensitivity and resistance to small molecule kinase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with unresectable or metastatic non-small cell lung cancer (NSCLC) and who fulfill the following eligibility criteria will be considered eligible for this study.

* Patient must have previously received treatment with small molecule kinase inhibitors targeting at least, in part, EGFR patients may have received other treatments since treatment with small molecule kinase inhibitors including radiation or chemotherapy)
* Development of disease progression while actively receiving tyrosine kinase inhibitor
* Signed informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unresectable or metastatic non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2004-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To compare EGFR gene sequence in patients upon relapse with EGFR gene sequence prior to treatment with small molecule kinase inhibitors. | 2 years

SECONDARY OUTCOMES:
To identify novel mutations in the tyrosine kinase domain of EGFR in patients with acquired resistance to small molecule kinase inhibitors. | 2 years
To more precisely characterize the frequency and clinical implications of T790M in patients with acquired resistance to small molecule kinase inhibitors. | 2 years
To identify novel mechanisms of acquired resistance to EGFR small molecule kinase inhibitors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- [Derived] Oxnard GR, Arcila ME, Sima CS, Riely GJ, Chmielecki J, Kris MG, Pao W, Ladanyi M, Miller VA. Acquired resistance to EGFR tyrosine kinase inhibitors in EGFR-mutant lung cancer: distinct natural history of patients with tumors harboring the T790M mutation. Clin Cancer Res. 2011 Mar 15;17(6):1616-22. doi: 10.1158/1078-0432.CCR-10-2692. Epub 2010 Dec 6. PMID 21135146
- See also: Related Info — http://www.mskcc.org